CLINICAL TRIAL: NCT02940964
Title: Evaluation of Culture-specific Popular Music as a Mental Metronome for Cardiopulmonary Resuscitation: A Randomized Crossover Trial
Brief Title: Evaluation of Culture-specific Popular Music as a Mental Metronome for Cardiopulmonary Resuscitation
Acronym: COMSCPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016/2773
Record Dates: First submitted 2016-10-17; First posted 2016-10-21 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Cardiac Arrest; Out-of-hospital Cardiac Arrest
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COMSCPR first (Experimental): Group A will proceed to perform one cycle (two minutes) of COMSCPR. After taking a fifteen minute rest, participants will cross over to perform one cycle of the other method of CPR.
  Interventions: Behavioral: Count on me Singapore (COMS) CPR
- Standard CPR first (Active Comparator): Group A will proceed to perform one cycle (two minutes) of Standard CPR. After taking a fifteen minute rest, participants will cross over to perform one cycle of the other method of CPR.
  Interventions: Behavioral: Standard CPR

INTERVENTIONS:
Behavioral: Count on me Singapore (COMS) CPR — Using the song as a mental metronome to guide CPR.
  Other Names: COMSCPR
  Arms: COMSCPR first
Behavioral: Standard CPR — Standard CPR with "one-and-two-and-three...." counting
  Arms: Standard CPR first

SUMMARY:
Abstract

Introduction

Bystander cardiopulmonary resuscitation (CPR) can more than double the patient's chance of survival in Out-of-hospital cardiac arrest (OHCA). In Singapore, bystander CPR rate was low. Recent studies have proposed and validated the use of popular songs as aids in performing CPR. These songs may not be widely known when applied to a different population, and further, may lose popularity over time. "Count on me Singapore" (COMS) is believed to be known to over 90% of the Singapore population. Pilot data indicated that CPR performed using COMS as a mental metronome (COMSCPR) can achieve guideline-compliant rate of chest compression with lower fatigue level than CPR guided by the conventional "one-and-two-three-and" (Standard CPR). The investigators hypothesize that COMSCPR is non-inferior to Standard CPR in achieving guideline-compliant rate of chest compression.

Methodology

The investigators planned a prospective, randomized, crossover non-inferiority trial comparing COMS CPR and Standard CPR. 80 eligible volunteers will be recruited from a convenience sample of camp personnel from a military training camp. After a 15 minutes familiarization session, they will be randomized into two groups (A and B). Group A will proceed to perform one cycle (two minutes) of Standard CPR, while group B will proceed to perform one cycle of COMS CPR. participants will cross over to perform one cycle of the other method of CPR. After completing this second cycle, a survey form will be administered. The Laerdal SkillReporter will be used to measure the CPR performed. After a 7-14 days interval, participants will be recalled to attend a test scenario. Statistical analysis will be used to compare the two arms.

ELIGIBILITY:
Inclusion Criteria:

* All volunteers are eligible. This mimics a real world situation where any trained member of the public can provide bystander CPR.

Exclusion Criteria:

* Lack of informed consent
* Existing medical conditions that may cause danger to the participant (e.g. cardiac conditions or musculoskeletal injuries)
* Recent CPR course attended (within past one month)

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2016-11-23 (Actual)

PRIMARY OUTCOMES:
Average compression rate | Immediately after 2 min of CPR
  As read by Laerdal SkillReporter

SECONDARY OUTCOMES:
Average depth of compression | Immediately after 2 min of CPR
  As read by Laerdal SkillReporter
Number of incorrect hand placement alerts | Immediately after 2 min of CPR
  As read by Laerdal SkillReporter
Number of compressions with inadequate recoil | Immediately after 2 min of CPR
  As read by Laerdal SkillReporter
Fatigue level after a cycle of CPR of 2 minutes duration, on a 10-point scale | Immediately after completing both types of CPR (crossover) 2 minutes
  Survey on a 10-point scale
Satisfaction of CPR provider in terms of ease of learning, fatigue and overall effectiveness assessed with a Survey on a 5-point scale | Immediately after completing both types of CPR (crossover) 2 minutes
  Survey on a 5-point scale
Ability to retain compression rate using COMS CPR after a 7-14 day interval with no additional prompting in between | Between 7-14 days
  As read by Laerdal SkillReporter

IPD SHARING:
Plan to Share IPD: Undecided